CLINICAL TRIAL: NCT05354089
Title: A Phase I, Randomized, Observer-blinded, Placebo-controlled and Dose-escalation Clinical Trial to Evaluate the Safety and Preliminary Immunogenicity of a SARS-CoV-2 mRNA Vaccine (SYS6006) in Chinese Healthy Adults Aged 18 -59 Years.
Brief Title: A Study of SARS-CoV-2 mRNA Vaccine (SYS6006) in Chinese Healthy Adults Aged 18 -59 Years.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYS6006-001
Record Dates: First submitted 2022-04-28; First posted 2022-04-29 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccine group 1 (Experimental): 20 μg dose of SYS6006 vaccine IM, on day 0 and day 21.
  Interventions: Biological: 20 μg dose of SYS6006
- Vaccine group 2 (Experimental): 30 μg dose of SYS6006 vaccine IM, on day 0 and day 21.
  Interventions: Biological: 30 μg dose of SYS6006
- Placebo (Placebo Comparator): Placebo IM, on day 0 and day 21.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: 20 μg dose of SYS6006 — 20 μg dose of SYS6006 vaccine IM on day 0 and day 21.
  Arms: Vaccine group 1
Biological: 30 μg dose of SYS6006 — 30 μg dose of SYS6006 vaccine IM on day 0 and day 21.
  Arms: Vaccine group 2
Drug: Placebo — Placebo IM on day 0 and day 21.
  Arms: Placebo

SUMMARY:
This is a phase I, randomized, observer-blinded, placebo-controlled and dose-escalation clinical trial to evaluate the safety, tolerability, immunogenicity and immune persistence of SYS6006 (SARS-CoV-2 mRNA Vaccine) in 18-59 year old healthy population.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of the first dose of vaccine: 18 to 59 years;
2. Axillary body temperature is less than 37.3 degree centigrade on the day of enrollment;
3. Based on the medical history and relevant physical examination and laboratory examination results (normal or abnormal but no clinical significance), the investigator clinically determined that the patient was in good health;
4. Has independent judgment, and participate voluntarily and sign an informed consent form.

Exclusion Criteria:

1. Has a history of SARS-CoV or SARS-CoV-2 infection, or close contact with SARS-CoV-2 infected persons (nucleic acid test positive) or living abroad within 30 days before screening;
2. Positive SARS-CoV-2 antibody test;
3. Previous history of allergy to acetaminophen or vaccination(eg, acute allergic reaction, urticaria, dyspnea, angioneurotic edema, or abdominal pain);
4. Has a history of COVID-19 vaccination, or have received other inactivated or recombinant vaccines within 7 days, or received live attenuated vaccines within 14 days,before the first dose;
5. Has a medical history or family history of epilepsy, convulsions, neurological diseases and psychiatric diseases;
6. Is contraindicative for intramuscular injection，such as: diagnosed thrombocytopenia, any coagulation disorders, or receiving anticoagulant therapy;
7. Has known or suspected serious disorders judged by the Investigator, including but not limited to respiratory disorders (pulmonary failure, etc.), liver and kidney disorders, cardiovascular disorders (cardiac failure, severe hypertension, etc.), malignant tumors, infections or allergic skin disorders, HIV infection, or in the acute infection or chronic disease activity period (within 3 days before vaccination);
8. Has chronic diseases (such as Down syndrome, sickle cell anemia, neurological disorders and Guillain-Barre syndrome, excluding stably controlled diabetes/hypertension) that are not suitable for this study at the discretion of the Investigator;
9. Has known immunocompromised conditions diagnosed in hospital before enrollment, or functional aspleen or splenectomy caused by any condition;
10. For women of childbearing potential: positive pregnancy test, being in pregnancy or breastfeeding, or have a pregnancy plan within one year;men: whose spouses is of childbearing potential and has a pregnancy plan within 1 year;
11. Is participating in other clinical trials or plan to participate in other clinical trials during the study period;
12. Has received immune enhancement or immunosuppressive therapy within 3 months before the first dose of vaccine (continuous oral or instillation for more than 14 days); or received whole blood, plasma and immunoglobulin therapy within one month;
13. Is unlikely to adhere to the study procedures or keep appointments at the discretion of the investigators;or plan to permanently relocate before the end of study; or plan to leave the resident location for a long time at the scheduled visit; or has any other conditions that are inappropriate for participation for this study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events, including solicited and unsolicited events | From the first dose through 30 days following the second dose.
adverse events associated with the study intervention | From the first dose through 30 days following the second dose.

SECONDARY OUTCOMES:
Geometric mean titer (GMT), geometric mean increase (GMI) and seroconversion rate (SCR) of anti-SARS-CoV-2 antibody (specific IgG antibody and neutralizing antibody) | 14 days after the first dose; 7 days, 14 days, 30 days, 90 days, 180 days and 360 days after the second dose
Serious adverse events (SAE) | from the first dose through 12 months after the second dose.
Adverse events of special interest (AESI) | from the first dose through 12 months after the second dose.
Laboratory test related adverse events | 4 days following each dose

CONTACTS AND LOCATIONS:
Overall Officials: Lanjuan Li, Principal Investigator — Shulan (Hangzhou) Hospital; Guiling Chen, Principal Investigator — Shulan (Hangzhou) Hospital; Xiang Lu, Principal Investigator — Sir Run Run Hosipital Nanjing Medical University; Yuwen Su, Principal Investigator — Sir Run Run Hosipital Nanjing Medical University
Locations (2):
- China (2):
  - Sir Run Run Hosipital Nanjing Medical University, Nanjing, Jiangsu
  - Shulan(hangzhou) Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No